CLINICAL TRIAL: NCT03963583
Title: Heart Failure Resilience Intervention for Caregivers (HEROIC)
Brief Title: Heart Failure Resilience Intervention for Caregivers
Acronym: HEROIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB00277814; 1K12HD085845 (NIH)
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Caregivers
Keywords: Heart Failure; Caregivers; Resilience; Preventive Health Behaviors
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEROIC Intervention Group (Experimental): This group will receive the HEROIC intervention.
  Interventions: Behavioral: HEROIC
- Waitlist Control Group (Experimental): The waitlisted group will receive usual care for caregivers for the first 12 weeks, which is normally limited to inclusion in some clinical assessment and teaching during patient visits. Waitlisted participants will receive monthly study postcards to encourage retention. After 12 weeks, they will begin the intervention.
  Interventions: Behavioral: HEROIC

INTERVENTIONS:
Behavioral: HEROIC — The HEROIC intervention will include individualized, nurse-led sessions focused on;
  1. a whole-person assessment including preventive health behaviors, personal goals, and purpose in life
  2. discussion of caregiving in the context of the caregiver's identified 'purpose' which supports meaning-making and provides rationale for goal-setting
  3. co-development of a plan to address caregiver goals to improve preventive health behaviors and/or reduce caregiver burden
  4. 'walking meetings' to model the importance of exercise while discussing incremental action plans to help caregivers achieve goals.

SUMMARY:
Heart failure (HF) patients with supportive caregivers have better physical health, emotional health, and quality of life. But caregivers have an increased risk of caregivers' own worsening health and often feel a sense of burden related to caregiving. However, caregivers receive very little support to balance caring for the patient with caring for themselves. Therefore, this research will provide a program for caregivers of advanced heart failure patients to build on the caregiver's strengths, sense of purpose, and set goals for healthy lifestyle changes. The investigators believe that caregivers who receive the program will have better quality of life, less sense of burden, and a healthier lifestyle.

DETAILED DESCRIPTION:
Aim 1) Develop the intervention through focus groups and human-centered design with key stakeholders with particular focus on race, gender and financial strain. Key stakeholders including patients, caregivers and healthcare providers will discuss prototypes and refine intervention components through human-centered design.

Aim 2) Refine intervention components through an open label pilot (N=5) of the intervention, followed by in-depth interviews. We will assess the salient features of the novel intervention components using mixed methods including examination of all quantitative measures and qualitative interviews to explore acceptability, participant/interventionist interactions, home environment factors, goal achievement and perceived value of intervention. Intervention components will be adapted for the trial based on results of aims 1 and 2.

Aim 3) Conduct a single-masked, waitlist control pilot trial of the HEROIC intervention (N=36). We hypothesize that caregivers who receive the intervention will show greater improvement in primary outcomes (preventive health behaviors, caregiver burden and QOL) and potential mechanisms (self-efficacy and biomarkers of resilience [interleukins 6 and 10]) than control caregivers.

Randomization: Caregivers will be randomized using a computer algorithm via REDCap to receive either: (1) intervention or (2) waitlist. Random assignment will be stratified by spousal vs non-spousal caregivers due to increased burden among non-spousal caregivers.

Waitlisted Control Group: The waitlisted group will receive usual care for caregivers for the first 16 weeks, which is normally limited to inclusion in some clinical assessment and teaching during patient visits. Waitlisted participants will receive monthly study postcards to encourage retention. After 16 weeks, they will begin the intervention.

Setting:

Aim 1: Key Stakeholder meetings will be held at the Johns Hopkins University School of Nursing, which is located within walking distance of the Heart Failure Bridge Clinic and supported by the Community Research Advisory Council.

Aims 2-3: Study visits will be conducted in the home of the caregiver.

Intervention Components

The intervention will be guided by the theory and evidence-based practices that have been successful in previous work. For the proposed study, every participant will receive each component of the intervention but interventionists will tailor content to each participant's goals. The investigators will focus on overall preventive health behaviors broadly categorized as physical activity, stress management, rest, healthy diet and appropriate healthcare utilization. As part of the intervention, the nurse and the caregiver will discuss preventive health categories. In this conversation, the caregiver will prioritize the preventive health categories that they would most like to address and then set goals towards them. Allowing the caregiver maximum control over this goal-setting, without placing additional burden on the caregiver is one aspect of increasing self-efficacy and person-centeredness. Because the intervention will allow participants to pick their own health goals, the investigators will measure goal attainment related to preventive health behaviors, rather than a standardized survey of predetermined preventive health behaviors.

Intervention Delivery/Study Visits

The intervention delivery characteristics will consist of an assessment-driven, tailored package of interventions delivered by a nurse interventionist. Nurse interventionists will be trained and equipped with education materials vetted by national organizations leading preventive health research such as the American Heart Association (Healthy for Good) and National Institute of Aging (Go4Life). The investigators propose an intervention incorporating 3 individualized, nurse-led, home-based sessions, with telephone check-ins and text reminders, according to participant preference. Baseline, 16 and 32-week data will be collected by interviewers masked to treatment assignment and without interventionist contact.

Interventional Protocol

The nurse will meet with the caregiver to perform the initial assessment in which the nurse will focus on preventive health behaviors and factors contributing to a sense of burden. To build rapport and model the importance of physical activity, the nurse will allow the caregiver to choose a short physical activity (ie. Walk around the block, 2 minutes of dancing etc). In this assessment, the nurse and the caregiver identify and prioritize goals, and make plans to achieve those goals. The nurse will provide the HEROIC Handbook, which will be developed following aim 1 and include evidence-based educational materials, contact information, and a calendar of sessions that the participant keeps for reference. In each session, the nurse assesses goal attainment, reinforces strategy use, reviews problem-solving, refines strategies (such as Go4Life physical activities and Healthy for Good materials), and provides education and resources to address future needs. Following the session, the nurse will find additional resources, tailored to each caregiver. In the final session, the nurse reviews the participants' strategies and helps to generalize them to other possible challenges or goals. Sessions will be spaced to encourage practicing new strategies independently after developing them together with the nurse. Although this intervention structure has been successful in work by the mentorship team, the investigators will adjust the timing and frequency of study visits based on feedback in phases 1 and 2. Bi-monthly meetings of the nurse with the site Research Coordinator and the principal investigator will ensure smooth communication, address challenges, supervision, and adherence to intervention fidelity.

ELIGIBILITY:
Inclusion criteria:

Aim 1 inclusion criteria:

* Patients with a HF hospitalization in the last year and their informal caregivers (inclusion criteria below), nurse practitioners, physicians and members of the multidisciplinary team rounds will be included in focus groups.

Aim 2 & 3 Inclusion:

* Caregivers of patients served by the HF Bridge Clinic will be included if

  1. the patient was hospitalized within 6 months
  2. the caregiver agrees to work on goals that increase preventive health behaviors and/or decrease burden
  3. caregivers live with the patient or visit them to provide care more than 3 times per week
  4. the caregiver is 50 years or older and e) the caregiver is the spouse/partner or child of the patient.

Exclusion criteria:

* Caregivers who

  1. themselves have a terminal diagnosis
  2. or are cognitively impaired based on Mini-Mental State Examination (MMSE) screening will be excluded as response to the intervention may vary in these groups.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Abshire Saylor, PhD, Principal Investigator — Johns Hopkins University School of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date
Access Criteria: The data may be used for any purpose. We will establish an online weblink.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 33 enrolled caregivers (participants): Withdrawn (n=10) , Lost to Follow-Up (n=2) , Determined not eligible (n=2), nineteen caregivers were randomized to the arms.
Period: Overall Study
Arm/Group | HEROIC Intervention Group | Waitlist Control Group
Started | 10 | 9
12-weeks | 8 | 9
Completed | 8 | 6
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HEROIC Intervention Group | Waitlist Control Group | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (10.7) | 55.9 (15.8) | 57.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 3 | 8
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Goal Attainment of Preventive Health Behaviors as Measured by the Goal Attainment Scale
Description: The Goal Attainment Scale is a self-reported attainment of goals implementing health-promoting behaviors, reported on a 5-point scale. Scores are converted to t-scores (0-100). 50 indicates the population mean with a standard deviation of 10. Higher scores indicate higher goal attainment.
Time Frame: Baseline, 12 and 24 weeks
Population: Participants with complete case data at each time point
Measure: Mean (Standard Deviation); unit: t-score
Arm/Group | HEROIC Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 8 | 6
t-score
  Baseline | 40 (0) | 40 (0)
  12 weeks | 57.5 (8.9) | 52.5 (13.9)
  24-weeks | 68 (4.5) | 51.7 (9.9)

2. Primary Outcome: Caregiver Burden as Assessed by the Oberst Caregiving Burden Scale
Description: Investigators will use the task difficulty and time caregiving subscales of the Oberst Caregiving Burden Scale. Both sub-scales include 15 likert scale items each. Scores range from 15-75 for the task difficulty and 15-75 for the time caregiving sub-scales. Higher scores indicate great task difficulty; higher scores indicate more time spent caregiving. Sub-scales are not combined in a total score.
Time Frame: Baseline, 12 and 24 weeks
Population: Participants with complete case data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HEROIC Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline - Difficulty | 50.2 (16.7) | 46.8 (17.8)
  12-weeks - Difficulty | 40.9 (18.3) | 43.0 (24.2)
  24-weeks - Difficulty | 34.4 (21.1) | 45.4 (27.9)
  Baseline - Time | 52.4 (13.1) | 49.3 (13.5)
  12-weeks - Time | 49.5 (13.5) | 51.6 (11.5)
  24-weeks - Time | 42.8 (21.3) | 57.4 (15.2)

3. Primary Outcome: Quality of Life as Assessed by the Neurological Quality of Life(Neuro-QOL)
Description: 9-Item Neurological Quality of Life (Neuro-QOL). Items are scored on a 1-5 range, with total summary score calculated range of 9-45. Higher scores indicate a more favorable quality of life.
Time Frame: Baseline, 12 and 24 weeks
Population: Participants with complete case data at each time point
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HEROIC Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline | 36.2 (6.2) | 34.4 (6.9)
  12-weeks | 37.3 (4.3) | 31.4 (8.0)
  24-weeks | 38.0 (5.5) | 33.5 (7.9)

4. Secondary Outcome: Self-Efficacy as Assessed by the Coping Self Efficacy Scale
Description: The coping self-efficacy scale has 13 items, each scored 0-10. Scores range from 0-130. Higher scores indicate higher coping self-efficacy.
Time Frame: Baseline, 12 and 24 weeks
Population: Participants with complete case data at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | HEROIC Intervention Group | Waitlist Control Group
Number analyzed (Participants) | 8 | 6
score on a scale
  Baseline | 92.1 (22.3) | 85.6 (26.1)
  12-weeks | 79.3 (34.1) | 71.0 (25.0)
  24-weeks | 98.5 (21.2) | 84.6 (30.8)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 24 weeks
Arm/Group | HEROIC Intervention Group | Waitlist Control Group
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-23): https://cdn.clinicaltrials.gov/large-docs/83/NCT03963583/Prot_SAP_000.pdf